CLINICAL TRIAL: NCT00364559
Title: Effect of Rosuvastatin on Outcome by NIHSS After Intracerebral Hemorrhage
Brief Title: Effect of Rosuvastatin in Intracerebral Hemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Humberto Tapia
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 29-09 ROICH
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Intracerebral Hemorrhage; Stroke
Keywords: intracerebral hemorrhage; statins; rosuvastatin; stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- B (Experimental): A, Active B, Historical Register
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg 10 days daily
  Other Names: Crestor

SUMMARY:
The purpose of this study is to determine whether rosuvastatin is effective in the management of acute phase of intracerebral hemorrhage and if it impact outcome by NIHSS.

DETAILED DESCRIPTION:
The intracerebral hemorrhage (ICH) is a frequent problem of health, with high morbid-mortality. In addition it originates expensive expenses in health care systems.

ICH produces damage by mass effect, then by biochemical ways which are activated and they carry to secondary damage. Many studies have been conducted for explaining secondary injury, now we know there are ischemic changes related maybe with changes in cerebral flow and metabolism, in addition to activate inflammatory ways. Many drugs and measures has been ineffective for getting best outcome, without success.

Statins or inhibitors of HMG CoA reductase are drugs used in dyslipidemia, frequently for reduction in LDL. Experimental and clinical studies in stroke and ICH have shown improvement in outcome. The toxicity related to statin is myopathy and hepatopathy, both with low incidence without fatal cases. Rosuvastatin has been postulated be the most powerful with longest life and toxicity similar to another statins.

We have designed this study to demonstrate if the administration of rosuvastatin in the first 24 hours and by 14 days has improvement in outcome.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women >16 and < 80 years with ICH and hospital attention in less 24 hours
* Confirmation by CT scan
* Acceptance by family

Exclusion Criteria:

* History of stroke
* History of neurological disease, head injury o psychiatric disorder with disability
* Glasgow less than 9
* Administration 24 hours before: fibrates, niacin, ciclosporin, azoles, macrolides, inhibitors of protease, nefazodone, verapamil, diltiazem, amiodarone.
* Use before hospital of: mannitol, barbiturates, corticosteroids, calcium antagonists
* Any lesion which needs surgery
* Allergy to drug used
* cerebral death
* Hepatic disease (Child B y C) or myopathy (or) history
* Management in other Hospital
* Pregnancy
* ICH major than 60 ml.
* hypothyroidism

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
NIHSSº | basal and discharge

SECONDARY OUTCOMES:
Survivor | within 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ildefonso Rodríguez-Leyva, Neurology, Study Director — Neurología, Hospital Central "Dr. ignacio Morones Prieto"; Humberto Tapia-Perez, MD, Principal Investigator — Facultad de Medicina UASLP
Locations (1):
- Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Tapia-Perez H, Sanchez-Aguilar M, Torres-Corzo J, Rodriguez-Leyva I, Herrera-Gonzalez LB. [Statins and brain protection mechanisms]. Rev Neurol. 2007 Sep 16-30;45(6):359-64. Spanish. PMID 17899518
- [Background] Tapia-Perez H, Torres-Corzo J, Sanchez-Aguilar M, Gonzalez-Aguirre D, Rodriguez-Leyva I, Teniente-Sanchez AE, Gordillo-Moscoso A. [A clinical-epidemiological approximation to intracerebral hemorrhage in a Mexican hospital: analysis of factors associated to mortality]. Rev Neurol. 2008 Jan 16-31;46(2):67-72. Spanish. PMID 18247276
- [Result] Tapia-Perez H, Sanchez-Aguilar M, Torres-Corzo JG, Rodriguez-Leyva I, Gonzalez-Aguirre D, Gordillo-Moscoso A, Chalita-Williams C. Use of statins for the treatment of spontaneous intracerebral hemorrhage: results of a pilot study. Cent Eur Neurosurg. 2009 Feb;70(1):15-20. doi: 10.1055/s-0028-1082064. Epub 2009 Feb 5. PMID 19197830